CLINICAL TRIAL: NCT03654625
Title: Development of a Scientifically-Informed Written Exposure Procedure (The SCRIPTS Study)
Brief Title: Development of a Scientifically Informed Written Exposure Procedure (The SCRIPTS Study)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Ministry of Research, Innovation and Science, Ontario (Other)
Responsible Party: Principal Investigator, Naomi Koerner, Associate Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB 2018-094
Record Dates: First submitted 2018-08-11; First posted 2018-08-31 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Excessive Worry
Keywords: Worry; Anxiety; Generalized Anxiety Disorder; Written Exposure
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: Baseline (pre-intervention) outcome measures will be completed at the first visit to the lab at Ryerson University. Participants will then be randomly assigned to one of the following conditions: (1) standard written exposure, (2) enhanced written exposure or (3) neutral writing. All participants will write at the lab for 30 minutes on each of 4 days. The 4 writing sessions will be spaced and take place within a 2-week period. During the 2-week intervention period and the three days following the intervention period, participants will track their worry and mood twice per day. With the exception of the Modified Behavioural Avoidance Test, which will only be assessed at pre-intervention and 1 month follow-up , all other outcomes will be reassessed at post-intervention, 1-week and 1-month follow-up. An additional assessment of excessive worry will occur at mid-intervention, and additional assessments of Perceived Probability, Cost and Coping Questions will occur at each writing session.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Written Exposure (Experimental): Four writing sessions at the laboratory
  Interventions: Behavioral: Standard Written Exposure
- Enhanced Written Exposure (Experimental): Four writing sessions at the laboratory
  Interventions: Behavioral: Enhanced Written Exposure
- Control Condition (Placebo Comparator): Four writing sessions at the laboratory
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Standard Written Exposure — Four spaced, 30-minute sessions occurring within a period of 2 weeks. Participants write a narrative about their worst worry.
  Arms: Standard Written Exposure
Behavioral: Enhanced Written Exposure — Four spaced, 30-minute sessions occurring within a period of 2 weeks. Participants write a narrative about their worst worry and rescript it.
  Arms: Enhanced Written Exposure
Behavioral: Control Condition — Four spaced, 30-minute sessions occurring within a period of 2 weeks. At each session, participants write a narrative about a neutral topic.
  Arms: Control Condition

SUMMARY:
Generalized anxiety disorder (GAD) is characterized by excessive and uncontrollable worry and anxiety. When people with GAD worry, they tend to think about problems and feared situations in a vague way. Preliminary research suggests that writing about feared situations in a structured and detailed fashion may help with worry. In this experiment, the investigators are looking to improve the writing intervention. The investigators are testing the immediate and short-term effects of a new writing intervention.

DETAILED DESCRIPTION:
Generalized anxiety disorder (GAD) is characterized by excessive and uncontrollable worry and anxiety about bad things that may happen in the future. When people with GAD worry, they tend to think about the situations they fear in a vague way. Preliminary research suggests that writing repeatedly about one's fears in a structured and detailed way may help worry. In the present experiment, the investigators are comparing three structured writing interventions and testing their immediate and short-term effects on worry, and worry-related features.

Potential participants will be asked to complete a telephone screen. Those who meet eligibility criteria will be invited to the laboratory at Ryerson University. After completing pre-intervention outcome measures, participants will be randomly assigned to one of three writing interventions: (1) standard written exposure, (2) enhanced written exposure, or (3) neutral writing. All participants will write for 30 minutes on each of 4 days. The 4 sessions of writing will be spaced and will take place within a period of 2 weeks. Excessive worry will be assessed at pre-intervention, mid-intervention, post-intervention, 1-week follow-up and 1 month follow-up. With the exception of the Modified Behavioural Avoidance Test, which will only be assessed at pre-intervention and 1 month follow-up, all other outcomes will be assessed at pre-intervention, and at post-intervention, 1-week follow-up and 1 month follow-up. Additional assessments of Perceived Probability, Cost and Coping Questions will occur at each writing session.

During the 2-week intervention period and the three days following the intervention period, all participants will also track their worry and mood twice per day.

The present experiment will provide answers to important questions about the therapeutic potential of writing interventions for excessive worry.

ELIGIBILITY:
Inclusion Criteria:

* Score of 56 or higher on the Penn State Worry Questionnaire.
* Endorsement of Generalized Anxiety Disorder as per the DSM-5 description (American Psychiatric Association, 2013).

Exclusion Criteria:

* Clinically significant suicidal ideation, intent, or plan
* Past or current history of psychosis or mania, or substance use disorder over the past 12 months
* Current psychological treatment or counseling unless this treatment is infrequent (once monthly or less) or the participant has been receiving consistent weekly treatment for at least 12 weeks and still meets all other eligibility criteria
* Psychotropic medication with a change in dose in the past 12 weeks. If they have recently discontinued a psychotropic medication, they will be included if it has been at least 1 month since discontinuation, or 3 months if they had been taking fluoxetine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2018-09-07 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported past-week worry as measured by the Penn State Worry Questionnaire-Past Week Version | Administered before the intervention on day 1 (pre-intervention), within week 2 of the intervention (at writing session 3), post-intervention (3 days after writing session 4), 1-week follow-up and 1-month follow-up.
  Self-report measure assessing the degree of excessive worry experienced over the past week. Fifteen items are summed to create a total score. Scores range from 0 to 90, with greater scores indicating a greater degree of worry.

SECONDARY OUTCOMES:
Self-reported generalized anxiety disorder symptoms as measured by the Generalized Anxiety Disorder Questionnaire for the Diagnostic and Statistical Manual of Mental Disorders (DSM) IV. | Administered before the intervention on day 1 (pre-intervention), post-intervention (3 days after writing session 4), 1-week follow-up, and 1-month follow-up.
  Self-report measure of GAD symptoms. Fourteen items are summed to create a total score. Total scores range from 0 to 12, with greater scores indicating greater GAD symptom severity.
Self-reported cognitive avoidance as measured by the Cognitive Avoidance Questionnaire | Administered before the intervention on day 1 (pre-intervention), post-intervention (3 days after writing session 4), 1-week follow-up, and 1-month follow-up.
  Self-report measure of the tendency to engage in various cognitive avoidance strategies. Twenty-five items are summed to create a total score. Total scores range from 25 to 125, with higher scores indicating greater cognitive avoidance.
Self-reported attitudes towards problems as measured by the Negative Problem Orientation Questionnaire | Administered before the intervention on day 1 (pre-intervention), post-intervention (3 days after writing session 4), 1-week follow-up, and 1-month follow-up.
  Self-report measure of attitudes towards problems. Twelve items are summed to create a total score. Total scores range from 12 to 60, with higher scores indicating greater negative attitudes towards problems.
Self-reported fear of emotions as measured by the Affective Control Scale | Administered before the intervention on day 1 (pre-intervention), post-intervention (3 days after writing session 4), 1-week follow-up, and 1-month follow-up.
  Self-report measure of fear of emotions and attempts to control emotional experience. The scale contains 42 items divided into four subscales for distinct emotions: anxiety; depression; anger; positive emotion. Total scores range from 42 to 294; subscale scores range from 13 to 91, with higher scores indicating a greater fear of emotions.
Self-reported perceptions of shame as measured by the Shame-Aversive Reactions Questionnaire | Administered before the intervention on day 1 (pre-intervention), post-intervention (3 days after writing session 4), 1-week follow-up, and 1-month follow-up.
  Self-report measure of perception of shame as an undesirable and painful emotion. Fourteen items are summed to create a total score. Total scores range from 14 to 98, with higher scores indicating higher levels of shame aversion.
Self-reported maladaptive beliefs as measured by the Early Maladaptive Schema Questionnaire - Research version | Administered before the intervention on day 1 (pre-intervention), post-intervention (3 days after writing session 4), 1-week follow-up, and 1-month follow-up.
  Self-report measure of stable maladaptive beliefs. The scale contains 75 items divided into fifteen subscales for distinct maladaptive beliefs. Subscale scores range from 0 to 15, with higher scores indicating greater maladaptive beliefs.
Self-reported worry-related behaviours as measured by the Worry Behaviours Inventory | Administered before the intervention on day 1 (pre-intervention), post-intervention (3 days after writing session 4), 1-week follow-up, and 1-month follow-up.
  Self-report measure of worry-related behaviours. Ten items are summed to create a total score. Total scores range from 0 to 40, with higher scores indicating greater engagement in avoidant behaviors that are associated with worry.
Self-reported mastery as measured by the Self-Mastery scale | Administered before the intervention on day 1 (pre-intervention), post-intervention (3 days after writing session 4), 1-week follow-up, and 1-month follow-up.
  Self-report measure that assesses the extent to which an individual perceives a sense of personal control or mastery over life outcomes. Seven items are summed to create a total score. Total scores range from 7 to 49, with higher scores indicating greater personal control or mastery.
Self-reported Perceived probability, cost and coping as measured by Perceived Probability, Cost and Coping questions | Administered before the intervention on day 1, within week 1 of the intervention (at writing session 2), within week 2 of the intervention (writing sessions 3 and 4), post-intervention (3 days after writing session 4), and 1-week and 1-month follow-up.
  Self-report measure of perceptions of probability and costliness of, and ability to cope with one's feared scenario. Three distinct questions assess each of the following perceptions related to feared scenarios: 1) Probability, 2) Cost and 3) Coping. Perceived probability scores range from 0 to 6 with higher scores indicating greater perceived likelihood of worst fears coming true. Perceived costliness scores range from 0 to 6, with higher scores indicating greater perceived costliness of worst fears. Perceived coping scores range from 0 to 6, with greater scores indicating greater ability to cope.
Fear and avoidance related to worst case scenario as measured by the Modified Behavioural Avoidance Test | Administered before the intervention on day 1 (pre-intervention) and 1-month follow-up.
  Participants are asked to hold a mental image in mind of their hypothetical worst case scenario and rate their level of fear from 0 (no fear at all) to 10 (the most fear), and desire to avoid the mental image from 0 (no desire to avoid imagining) to 10 (the highest possible desire to avoid imagining).
Self-reported depression, anxiety and stress as measured by the Depression, Anxiety and Stress Scale | Administered before the intervention on day 1 (pre-intervention), post-intervention (3 days after writing session 4), 1-week follow-up, and 1-month follow-up.
  Self-report measure that assesses depression, anxiety and stress symptoms over the past week. The scale contains 21 items, divided into three subscales: 1) Depression, 2) Anxiety and 3) Stress. Scores on the subscales range from 0 to 42, with higher scores indicating greater severity of depression, anxiety and stress.
Daily Worry and Emotion Questions | During the two-week intervention period and for three days following the intervention period, all participants are asked to respond to questions about their worry and emotions twice per day (morning and evening) using an online diary.
  A daily self-report measure of (1) emotions, (2) worry controllability, (3) worry intensity and (4) worry duration.
  Scores for the first three items range from 0 to 8, with higher scores indicating greater degree of emotions, worry intensity, and difficulty controlling worry. Worry duration is reported in minutes, with greater numbers indicating longer time spent worrying.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Koerner, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- Ryerson University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Results of the study will be disseminated via conference presentations, journal publications, and through our lab website. Upon request, anonymized aggregate participant data may be made available to a publishing journal or individual research group. Individual research groups interested in accessing anonymized data will be required to submit a proposal detailing their intended use of the data. Their qualifications will be reviewed based on their proposal and curricula vitae (CVs). Individual research groups approved for access will be required to agree to not attempt to re-identify participants, not further distribute data, and not use the data for purposes other than specified in their original proposal. No individual data will be shared.

REFERENCES:
- [Background] Fracalanza K, Koerner N, Antony MM. Testing a procedural variant of written imaginal exposure for generalized anxiety disorder. J Anxiety Disord. 2014 Aug;28(6):559-69. doi: 10.1016/j.janxdis.2014.05.011. Epub 2014 Jun 14. PMID 24983797
- See also: Lab website — https://psychlabs.ryerson.ca/caplab/